CLINICAL TRIAL: NCT02496585
Title: Phase II Double-Blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of Nintedanib (BIBF 1120) + Prednisone Taper in Patients With Radiation Pneumonitis
Brief Title: Study to Evaluate the Efficacy and Safety of Nintedanib (BIBF 1120) + Prednisone Taper in Patients With Radiation Pneumonitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-167
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer; Lung Metastases
Keywords: Nintedanib (BIBF 1120); Prednisone; Radiation Pneumonitis
MeSH Terms: conditions — Lung Neoplasms; Radiation Pneumonitis | interventions — nintedanib; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nintedanib + Prednisone (Experimental): The initial dose of nintedanib will be 150mg two times per day orally according to study protocol. Nintedanib will be taken for 12 weeks. Patients will be given a prednisone taper (40mg prednisone daily for 2 weeks, followed by a strict dose taper of 10mg every 2 weeks for 4 weeks, followed by 10mg for one week and 5mg for one week, for a total duration on prednisone of 8 weeks).
  Interventions: Drug: Nintedanib; Drug: Prednisone
- Placebo + Prednisone (Experimental): Placebo will be taken for 12 weeks. Patients will be given a prednisone taper (40mg prednisone daily for 2 weeks, followed by a strict dose taper of 10mg every 2 weeks for 4 weeks, followed by 10mg for one week and 5mg for one week, for a total duration on prednisone of 8 weeks).
  Interventions: Drug: Prednisone; Other: Placebo

INTERVENTIONS:
Drug: Nintedanib
  Other Names: BIBF 1120
  Arms: Nintedanib + Prednisone
Drug: Prednisone
Other: Placebo
  Arms: Placebo + Prednisone

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the drug nintedanib in combination with steroids, has on the lungs. Furthermore, such treatments' side effects will be studied together with quality of life. In addition, the investigators would like to determine whether they can find markers in the blood which predict worsening lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven primary thoracic or breast malignancy, lymphoma or lung metastases (which are not required to be biopsy-proven) treated with definitive intent at MSK
* Prior treatment with thoracic radiotherapy completed >4 weeks and ≤ 9 months prior to enrollment
* Radiographic evidence of radiation pneumonitis on a CT scan of the chest with or without contrast
* Newly diagnosed clinical grade 2 or higher radiation pneumonitis according to CTCAE version 4.0 criteria
* Age≥18 years
* KPS > 70%
* Reduction of any acute toxicity from radiation treatment to grade 1
* Written informed consent signed prior to entry into the study

Exclusion Criteria:

* Current oral steroid use > 4 weeks prior to registration
* Ongoing treatment with radiotherapy to thorax, cytotoxic or biological therapies for this malignancy, except the following therapies which are permitted: Pembrolizumab, Nivolumab, Afatinib and all hormonal therapies.
* Mean esophageal radiation dose >45 Gy
* Diagnosis of diffuse radiation pneumonitis
* Untreated or symptomatic brain metastases or leptomeningeal disease
* Liver metastases
* Other active malignancies requiring oncologic treatment (Note: non-melanoma skin cancer, superficial bladder cancer etc. are eligible)
* Radiographic evidence of cavitary or necrotic tumor and local invasion of major blood vessels
* Active chronic Hepatitis C and/or B infection
* Gastrointestinal disorders that would interfere with drug absorption
* AST > 1.5 x ULN, ALT>1.5 x ULN and Bilirubin > 1.5 x ULN
* ≥ Grade 2 proteinuria, creatinine >1.5x ULN or GFR <45 ml/min
* Other investigational therapy received within 8 weeks prior to screening visit
* Pregnant women or women who are breast feeding or of child bearing potential not using a highly effective method of birth control for at least one month prior to enrollment1
* Sexually active males not committing to birth control during the course of the study (except if their partner is not of childbearing potential)
* Conditions that may affect the patient's ability to participate in this trial, e.g. known or suspected active alcohol or drug abuse
* Inherited predisposition to bleeding or thrombosis, INR >2, PT and PTT >1.5x ULN
* History of bleeding disorders or thrombotic events, e.g. hemorrhagic or thrombotic events within 12 months, clinically significant or tumor-related hemoptysis, active gastrointestinal bleeding or ulcers or major injuries or surgery
* ANC < 1.5 K/mcL, Platelets < 100 K/mcL, Hemoglobin < 9.0 g/dl
* Concomitant treatment with any of the following drugs: azathioprine, cyclophosphamide, cyclosporine, pirfenidone, full dose anticoagulation (vitamin K antagonists, dabigatran, heparin, etc.), fibrinolysis and high dose anti-platelet therapy (ex. Plavix 150mg)^2 Myocardial infarction or unstable angina within 6 or 1 month of starting nintedanib treatment, respectively
* Known inherited predisposition to thrombosis
* Patient with a history of a thrombotic event within 12 months of starting nintedanib treatment
* Known predisposition to bleeding
* Patients with severe hepatic impairment
* History of a gastrointestinal perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Moore, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Brigham and Women's Hospital (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania
  - MD ANDERSON CANCER CENTER (Data Collection Only), Houston, Texas
  - Myriad Genetic Laboratory (Data or Specimen Analysis Only), Salt Lake City, Utah

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib + Prednisone: The initial dose of nintedanib will be 150mg two times per day orally according to study protocol. Nintedanib will be taken for 12 weeks. Patients will be given a prednisone taper (40mg prednisone daily for 2 weeks, followed by a strict dose taper of 10mg every 2 weeks for 4 weeks, followed by 10mg for one week and 5mg for one week, for a total duration on prednisone of 8 weeks).
  Nintedanib
  Prednisone
- Placebo + Prednisone: Placebo will be taken for 12 weeks. Patients will be given a prednisone taper (40mg prednisone daily for 2 weeks, followed by a strict dose taper of 10mg every 2 weeks for 4 weeks, followed by 10mg for one week and 5mg for one week, for a total duration on prednisone of 8 weeks).
  Prednisone
  Placebo
Period: Overall Study
Arm/Group | Nintedanib + Prednisone | Placebo + Prednisone
Started | 19 | 15
Completed | 9 | 12
Not Completed | 10 | 3
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Progression of Malignancy | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib + Prednisone | Placebo + Prednisone | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Continuous [Mean (Full Range); unit: years] | 72 [58 to 80] | 70 [47 to 86] | 71 [47 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 8 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Are Free From Pulmonary Exacerbations
Description: An acute exacerbation will be defined as (all criteria must be met):
  1. Unexplained worsening or development of cough, dyspnea, hypoxia, or pneumonitis lasting more than 4 days
  2. New or worsening diffuse pulmonary infiltrates on chest CT (with or without contrast) or new high resolution CT parenchymal abnormalities without significant pneumothorax or pleural effusion
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percental of participants
Arm/Group | Nintedanib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 18 | 12
percental of participants | 72 [54 to 96] | 40 [20 to 82]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Nintedanib + Prednisone | Placebo + Prednisone
All-Cause Mortality (participants affected / at risk) | 8/18 | 3/12
Serious Adverse Events (participants affected / at risk) | 7/18 | 1/12
Other Adverse Events (participants affected / at risk) | 18/18 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib + Prednisone (N=18) | Placebo + Prednisone (N=12)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infection (Infections and infestations) | 3 | 0
Pain (General disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shingles (Infections and infestations) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib + Prednisone (N=18) | Placebo + Prednisone (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Blurred vision (Eye disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 11 | 5
Dizziness (Nervous system disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dry throat (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Edema limbs (General disorders) | 1 | 1
Elevated liver enzymes (Investigations) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 1
Eyelid function disorder (Eye disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 9 | 8
Fever (General disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 2
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hot flashes (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Influenza Type A (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Irritability (Psychiatric disorders) | 0 | 1
Left mid back mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liver enzyme elevations (Metabolism and nutrition disorders) | 1 | 0
Lung infection (Infections and infestations) | 3 | 0
Lymphocyte count decreased (Investigations) | 2 | 1
Malaise (General disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Parenchymal changes (Injury, poisoning and procedural complications) | 3 | 2
Paresthesia (Nervous system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 3
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Polyphagia (Gastrointestinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Shingles (Infections and infestations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Spasticity (Nervous system disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Tremor (Nervous system disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
White blood cell decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT02496585/Prot_SAP_000.pdf